CLINICAL TRIAL: NCT05448157
Title: 68Ga-DOTATOC Radio-Guided Surgery With β-Probe in GEP-NET
Acronym: RGS-GEP-NET
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: European Institute of Oncology (Other)
Responsible Party: Principal Investigator, Emilo Bertani, Director - surgeon, European Institute of Oncology
Other Study IDs: IEO 1740
Record Dates: First submitted 2022-07-01; First posted 2022-07-07 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Neuroendocrine Tumor Carcinoid; Neuroendocrine Tumor of Pancreas; Gep Net
MeSH Terms: conditions — Carcinoid Tumor; Adenoma, Islet Cell; Gastro-enteropancreatic neuroendocrine tumor

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — small bowel and mesenteric lymph-nodes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In gastro-entero-pancreatic neuroendocrine tumors (GEP-NETs), radical surgery provides good long-term outcome and low recurrence rates. In GEP-NETs the actual surgical planning is established on the ground of preoperative morphology images (CT scan), and functional imaging using CT/PET with 68Ga-DOTA-TOC, since the high expression of somatostatin receptors (SSR) of these tumors. RGS in GEP-NETs, mainly with gamma-probes, has been not widely accepted since the low rates of sensitivity and, in particular, specificity, in discriminating tumoral/ non tumoral tissue and background ratio. This is a relevant issue in particular in detecting metastatic lymph-nodes both for small-intestine neuroendocrine tumors (SI-NETs) and pancreatic neuroendocrine tumors (Pan-NETs), where the presence of lymph-node metastases has been associated with worse long-term outcome. At present, it is not possible to distinguish whether a small lymph-node is site of metastases or not without performing frozen sections. In a previous study ex-vivo from European Institute of Oncology SI-NET presented a high uptake of a beta-emitting radiotracer, 90Y-DOTA-TOC. Five SI-NET showing SSR positivity at PET with 68Ga DOTA-TOC received 5 mCi of 90Y-DOTA-TOC the day before surgery. All the tumor samples showed high counts of radioactivity with a sensitivity of 96% and a specificity of 100%. These results allowed the investigators to develop a probe, which is now approved for in-vivo employment within the operating theatre. The objective of the present study is to verify in-vivo within the abdominal cavity the capability of the probe to detect 68-Ga activity within tumoral tissue thus favouring radical surgery and avoiding unnecessary demolition, in the near future. However, in the present protocol the entity of surgery will not be modified by intraoperative findings of the probe. It is reasonable to assume that results from 68Ga-DOTA-TOC might be comparable to 90Y-DOTA-TOC as radiotracer, and the detection efficacy of the probe for 68Ga could be not inferior compared to the isotope 90Y. However, while 90Y-DOTA-TOC is used as investigational drug for therapy purposes only within clinical research protocol, 68Ga-DOTA-TOC is a diagnostic radiotracer broadly used in day-to-day clinical practice since many years. Furthermore, the administration of 68Ga-DOTA-TOC can be directly injected in surgery room and thus does not require patients' admission the day before surgery.

DETAILED DESCRIPTION:
Radical surgery is one of the most important way of treatment for solid tumors. In gastro-entero-pancreatic neuroendocrine tumors (GEP-NETs), it provides good long-term outcome and low recurrence rates. For breast cancer radio-guided surgery (RGS), using gamma radiations, is a well standardised methods because it aids to remove non-palpable lesions. In GEP-NETs the actual surgical planning is established on the ground of preoperative morphology images (CT scan), and functional imaging using CT/PET with 68Ga-DOTA-TOC, since the high expression of somatostatin receptors (SSR) of these tumors. RGS in GEP-NETs, mainly with gamma-probes, has been not widely accepted since the low rates of sensitivity and, in particular, specificity, in discriminating tumoral/ non tumoral tissue and background ratio. This is a relevant issue in particular in detecting metastatic lymph-nodes both for small-intestine neuroendocrine tumors (SI-NETs) and pancreatic neuroendocrine tumors (Pan-NETs), where the presence of lymph-node metastases has been associated with worse long-term outcome. At present, it is not possible to distinguish whether a small lymph-node is site of metastases or not without performing frozen sections. In a previous study ex-vivo from our Institute SI-NET presented a high uptake of a beta-emitting radiotracer, 90Y-DOTA-TOC. Five SI-NET showing SSR positivity at PET with 68Ga DOTA-TOC received 5 mCi of 90Y-DOTA-TOC the day before surgery. All the tumor samples showed high counts of radioactivity with a sensitivity of 96% and a specificity of 100%. These results allowed us to develop a probe, which is now approved for in-vivo employment within the operating theatre. The objective of this study is to verify in-vivo within the abdominal cavity the capability of the probe to detect 68-Ga activity within tumoral tissue thus favouring radical surgery and avoiding unnecessary demolition, in the near future. However, in the present protocol the entity of surgery will not be modified by intraoperative findings of the probe. It is reasonable to assume that results from 68Ga-DOTA-TOC might be comparable to 90Y-DOTA-TOC as radiotracer, and the detection efficacy of the probe for 68Ga could be not inferior compared to the isotope 90Y. However, while 90Y-DOTA-TOC is used as investigational drug for therapy purposes only within clinical research protocol, 68Ga-DOTA-TOC is a diagnostic radiotracer broadly used in day-to-day clinical practice since many years. Furthermore, the administration of 68Ga-DOTA-TOC can be directly injected in surgery room and thus does not require patients' admission the day before surgery.

The Primary objectives are to evaluate the diagnostic accuracy of the combined approach with β-probe and 68Ga-68 DOTA-TOC PET/CT in the correct identification of primary tumor and lymph-node metastases, patients with gastro-entero-pancreatic neuroendocrine tumors (GEP-NET) undergoing surgery. The histopathological analysis of the surgical specimens will be considered the standard of reference and diagnostic accuracy will be evaluated in terms of sensitivity and specificity.

The secondary objectives are:

* the identification of the most appropriate tumor-to-background ratio (TBR) able to correctly locate the signal emitted by DOTA-TOC-positive tumors or lymph nodes compared with the signal derived by the background rumor.
* safety and toxicity analysis regarding the intraoperative application of the β-probe.
* the comparison between the signal detected by the β-probe and 68Ga-DOTA-TOC PET/CT images.
* the correlation of the signal detected by the β-probe with the DOTA-TOC expression (DOTA-TOC staining) in tumors AND lymph node metastases assessed by immuno-histochemical analysis on the surgical specimens

The pathology assessment will be assessed with Immune-histo-chemical (IHC) analysis performed on surgical specimens obtained during surgery to assess the presence of neuroendocrine tumor localizations

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven GEP-NET
* Patients undergoing primary tumor and/or lymph-node dissection after discussion at IEO NET tumor board
* 68Ga-DOTA-TOC PET/CT performed within 12 weeks prior to surgery
* DOTA-TOC positive tumors 68Ga-DOTA-TOC PET/CT
* Age >18 years old
* Willing to sign informed consent

Exclusion Criteria:

* Patient unfit for surgery
* Patients negative to 68Ga-DOTA-TOC PET/CT
* Unable to tolerate PET scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with GEP-NET undergoing surgery who performed 68Ga-DOTA-TOC PET/CT per clinical routine practice will be considered suitable for enrollment in case of PET/CT positivity. Both metastatic and non-metastatic patients will be eligible
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-12-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the diagnostic efficacy and the safety of the combined approach with β-probe and 68Ga-DOTA-TOC PET/CT in the correct identification of primary tumor and lymph node metastases, in patients with GEP-NETs candidates to surgery | During surgical procedure
  The histopathological analysis of the surgical specimens will be considered the standard of reference and diagnostic efficacy will be evaluated in terms of sensitivity, specificity and positive predictive value (PPV). The radiation protection considerations are related to administering 68Ga-DOTA-TOC-PET/CT to enable radio-guided surgery. The day of surgery, the patients enrolled will receive 1.1 MBq/Kg, 60-90 minutes prior to surgery. The activity has been calculated considering preliminary in humans' data recently published by Collamati at al. Moreover, on the basis of the results of the first patients, the activity to be administered could be further reduced, considering that the beta probe detection will be performed approximately 1 hour after administration and not after 3 hours as reported in the reference. In any case, for radiation protection purposes only, it will be assumed that all 12 patients will be given an activity of 1.1 MBq/Kg.

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Bertani, Principal Investigator — IRCCS Istituto Europeo di Oncologia S.r.l.
Locations (1):
- IRCCS Istituto Europeo di Oncologia S.r.l., Milan, Italy

REFERENCES:
- [Derived] Bertani E, Mattana F, Collamati F, Ferrari ME, Bagnardi V, Frassoni S, Pisa E, Mirabelli R, Morganti S, Fazio N, Fumagalli Romario U, Ceci F. Radio-Guided Surgery with a New-Generation beta-Probe for Radiolabeled Somatostatin Analog, in Patients with Small Intestinal Neuroendocrine Tumors. Ann Surg Oncol. 2024 Jul;31(7):4189-4196. doi: 10.1245/s10434-024-15277-x. Epub 2024 Apr 23. PMID 38652200